CLINICAL TRIAL: NCT05685654
Title: Prospective Study to Validate the Clinical Accuracy of the Norbert Device to Measure Oxygen Saturation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Norbert Health (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: NCP-0003
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Healthy; Hypoxia
Keywords: medical device; validation; hypoxia; SpO2; oxygen saturation; Norbert Device; Norbert Health
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Norbert Device — The Norbert Device (ND) is a contactless, noninvasive device that provides measurements of body temperature, oxygen saturation (SpO2), and pulse rate.

SUMMARY:
The purpose of this study is to evaluate the SpO2 accuracy and performance of the Norbert Device during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-oximetry for SpO2 validation.

DETAILED DESCRIPTION:
The study is a single center, prospective, non-randomized study to measure the accuracy of an investigational device compared to blood reference values. The design of the study will be conducted in accordance with the recommendations of ISO 80601-2-61:2011 Annex EE.2 Procedure for invasive laboratory testing on healthy volunteers. The purpose of this study is to evaluate the SpO2 accuracy and performance of the Norbert Device during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-oximetry for SpO2 validation. The end goal is to show the SpO2 accuracy performance of the Norbert Device. It is expected that the Accuracy Root Mean Square (Arms) performance of pulse oximeters will meet a specification of 3.5 or better in non-motion conditions for the range of 70-100% SaO2 thereby demonstrating an acceptable SpO2 accuracy performance specification.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female subjects between the ages of 18 to 50 years
* Completion of a health screening for a medical history by a licensed physician, nurse practitioner, or physician assistant
* Previously measured hemoglobin electrophoresis with normal result recorded in Duke Epic EHR
* Minimum weight 40kg; BMI within range 18.0 - 35.0
* Assigned American Society of Anesthesiologists (ASA) Physical Status 1 by Principal Investigator or delegate

Exclusion Criteria:

* Prior or known allergies to lidocaine (or similar pharmacologic agents, e.g., Novocain)
* Prior known severe allergies to medical grade adhesive/tape (Band-Aid)
* Taking any medication other than birth control
* Is currently participating in, or has recently participated in (discontinued within 30 days prior to the hypoxia procedure for this study) in an investigational interventional drug, device, or biologic study
* Has a negative Allen's Test to confirm non patency of the collateral artery
* Has made a whole blood donation or has had at least 450 ml of blood drawn within 8 weeks prior to the study procedure
* Is female with a positive urine pregnancy test, or is female and is unwilling to use effective birth control between the time of screening and study procedure or is breast feeding
* Has anemia
* Has heparin allergy
* Has a history of sickle cell trait or thalassemia [self-reported]
* Has a positive urine cotinine test or urine drug screen or oral ethanol test
* Has a room air saturation less than 95% by pulse oximetry
* Has a clinically significant abnormal EKG
* Has a COHb greater than 3%, or MetHb greater than 2%
* Students and Employees under the direct supervision of PI or Sub-I

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 15 healthy, adult volunteers, aged 18 - 50, will be enrolled. The subjects will be distributed across both genders as equally as practical and with a range of skin pigmentation.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
SpO2 root mean square accuracy of the Norbert Device | Up to 1 hour
  SpO2 root mean square accuracy will be calculated following FDA guidelines.
SpO2 bias of the Norbert Device | Up to 1 hour
  SpO2 bias calculation of the Norbert Device will follow the FDA guidelines for analyzing population mean bias, between-subject variance, and within-subject variance.
Bland-Altman plots with linear regression line and 95% upper and lower limits of agreement | Up to 1 hour
  A method comparison study will be analyzed with a Bland-Altman plot. This study will produce limits of agreement (LoA) and associated confidence intervals from the two measurements obtained on each subject. The conclusion that the two measurements are in agreement depends on whether the confidence intervals constructed from the data are within the boundaries set from the maximum allowable difference.

IPD SHARING:
Plan to Share IPD: No